CLINICAL TRIAL: NCT00838682
Title: Effect of High-dose Oral Rabeprazole on Recurrent Bleeding After the Endoscopic Treatment of Bleeding Peptic Ulcers
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated before the complete enrollment due to slow enrollment
Sponsor: The Catholic University of Korea (Other)
Collaborators: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: HiunSuk Chae, The Catholic University of Korea College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAB-KOR-18
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Results first posted 2010-09-24 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-08

CONDITIONS: Peptic Ulcer Hemorrhage
Keywords: peptic ulcer bleeding; rabeprazole; proton pump inhibitor
MeSH Terms: conditions — Peptic Ulcer Hemorrhage | interventions — Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- rabeprazole sodium (Experimental): Oral Rabeprazole 20 mg twice daily for 3 days. From Day 4, oral Rabeprazole 10 mg once daily for 6 weeks as maintenance therapy.
  Interventions: Drug: Rabeprazole
- Omeprazole (Active Comparator): Intravenous Omeprazole 80 mg as a bolus injection followed by continuous infusion at 8 mg per hour for 3 days. From Day 4, oral Rabeprazole 10 mg once daily for 6 weeks as maintenance therapy.
  Interventions: Drug: omeprazole sodium IV

INTERVENTIONS:
Drug: omeprazole sodium IV — Intravenous Omeprazole (brand name: Losec® injection 40 mg) 80 mg as a bolus injection followed by continuous infusion at 8 mg per hour for 3 days. From Day 4, oral Rabeprazole 10 mg once daily for 6 weeks as maintenance therapy.
  Other Names: Losec IV
  Arms: Omeprazole
Drug: Rabeprazole — Oral Rabeprazole 20 mg twice daily for 3 days. From Day 4, oral Rabeprazole 10 mg once daily for 6 weeks as maintenance therapy.
  Other Names: Pariet
  Arms: rabeprazole sodium

SUMMARY:
This study is conducted to compare and evaluate the effect of administering a high-dose intravenous proton pump inhibitors or high-dose oral Rabeprazole in preventing recurrent bleeding after the endoscopic treatment of bleeding peptic ulcers.

DETAILED DESCRIPTION:
0.1 % of hospitalized patients are attributed to upper gastrointestinal bleeding every year in the U.S. and Europe, among which peptic ulcer is the most common cause of upper gastrointestinal bleeding. Endoscopic hemostasis procedure in the management of bleeding due to peptic ulcers was safe as well as effective and lowered recurrent bleeding, surgery and mortality. Endoscopic treatment is widely used as an effective and safe method but it has disadvantages including the need for the endoscopy specialist and the likelihood of developing the complications such as perforation or recurrent bleeding although they rarely occur. Thus, less invasive medical treatments with fewer side effects have been continuously studied and among them, gastric acid inhibitors have been studied the most.Acid and pepsin inhibit platelet aggregation, activation of blood coagulation system, and fibrinogen polymerization. Blood clots already formed are digested by pepsin and the activity of pepsin is closely related to intragastric pH level. Therefore, it is known that an elevated intragastric pH facilitates hemostasis process, induces hemostasis by stabilizing hematoma and prevents recurrent bleeding. To suffice these conditions, it is reported that a potent gastric acid inhibitor is needed to maintain intragastric pH of 6 or higher.

For the treatment of bleeding peptic ulcers, the intravenous administration of a high-dose proton pump inhibitor after the initial endoscopic treatment has shown a decline in the frequency of recurrent bleeding as well as surgery. Recent studies reported that the use of oral proton pump inhibitor was effective under certain circumstances in the treatment of bleeding peptic ulcers. However, to date, no study has been conducted to compare the effect of a high-dose intravenous proton pump inhibitor with that of oral Rabeprazole after endoscopic treatment of bleeding peptic ulcers. Therefore, in this study, after administering a high-dose intravenous proton pump inhibitor or high-dose oral Rabeprazole in preventing recurrent bleeding following endoscopic treatment of bleeding peptic ulcers, we are going to compare the rate of recurrent bleeding between the two groups as well as to compare and evaluate the surgery rate, mortality rate and the number of days of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Bleeding peptic ulcer: Among patients suspected to have upper GI bleeding based on hematemesis or melena, those with peptic ulcers(Forrest I, IIa and IIb) in whom active bleeding, non-bleeding visible vessels and fresh blood clots are observed on upper GI endoscopy performed within 24 hours after the hospitalization
* patients who achieved primary hemostasis with endoscopic hemostasis procedure via upper GI endoscopy

Exclusion Criteria:

* Patients who refuse endoscopic procedure
* Patients with complications from gastric ulcer that require operative treatment prior to upper GI endoscopic treatment(e.g., gastric outlet obstruction, peptic ulcer perforation)
* Pregnancy
* Patients with serious concurrent diseases such as malignant tumors or end-stage diseases
* History of previous gastrectomy or vagotomy
* Known hypersensitivity to proton pump inhibitors
* Elderly patients
* Epilepsy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2006-04; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiun-Suk Chae, Professor, Principal Investigator — The Catholic University of Korea
Locations (2):
- South Korea (2):
  - Bucheon St. Mary's Hospital, Bucheon-si, Kyungkido
  - Uijeongbu St.Mary's Hospital, Uijeongbu-si, Kyungkido

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1. Location: Uijeongbu St. Mary's hospital and Bucheon St. Mary's hospital, The Catholic University of Korea
  2. Period: from April 1, 2006 to April 19, 2007 and from October 1, 2007 to December 31, 2008.
Pre-assignment Details: Patients who presented with overt or suspected upper gastrointestinal bleeding were eligible. These eligible patients were required to have an high-risk bleeding peptic ulcer on emergent endoscopy performed within 24 hours after the hospitalization. Among those, patients who achieved primary hemostasis with endoscopic hemostatic treatment.
Period: Overall Study
Arm/Group | Rabeprazole Sodium | Omeprazole
Started | 54 | 52
Completed | 29 | 33
Not Completed | 25 | 19
Not completed — Lost to Follow-up | 21 | 14
Not completed — detection of exclusion criteria | 4 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rabeprazole Sodium | Omeprazole | Total
Number analyzed (Participants) | 54 | 52 | 106
Age Continuous [Mean (Standard Deviation); unit: years] | 56.1 (16.2) | 57.1 (15.8) | 56.6 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 21
  Male | 46 | 39 | 85
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 54 | 52 | 106

OUTCOME MEASURES:

1. Primary Outcome: Rebleeding Within 3 Days
Time Frame: day 3
Population: intention to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Rabeprazole Sodium | Omeprazole
Number analyzed (Participants) | 54 | 52
participants | 2 | 1
Statistical Analysis 1: Comparison: Rabeprazole Sodium vs Omeprazole; Test type: Superiority or Other; p < 0.05, Fisher Exact

2. Secondary Outcome: Rebleeding After 3 Days
Description: Rebleeding after 3 days was assessed by checking the patients from day 3 to discharge and bleeding event or regular follow-up after discharge to week 6.
Time Frame: 6wk
Population: intention to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Rabeprazole Sodium | Omeprazole
Number analyzed (Participants) | 54 | 52
participants | 1 | 0
Statistical Analysis 1: Comparison: Rabeprazole Sodium vs Omeprazole; Test type: Superiority or Other; p < 0.05, Fisher Exact

3. Secondary Outcome: Surgery
Description: This sencodary endpoint "surgery" is the operation for bleeding control of peptic ulcer bleeding such as gastric or duodenal primary closure, and subtotal gastrectomy with/without vagotomy.
Time Frame: 6wk
Population: intention to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Rabeprazole Sodium | Omeprazole
Number analyzed (Participants) | 54 | 52
participants | 2 | 0
Statistical Analysis 1: Comparison: Rabeprazole Sodium vs Omeprazole; Test type: Superiority or Other; p < 0.05, Fisher Exact

4. Secondary Outcome: Death
Time Frame: 6wk
Population: intention to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Rabeprazole Sodium | Omeprazole
Number analyzed (Participants) | 54 | 52
participants | 1 | 0
Statistical Analysis 1: Comparison: Rabeprazole Sodium vs Omeprazole; Test type: Superiority or Other; p < 0.05, Fisher Exact

5. Other Pre Specified Outcome: Mean Units of Blood Transfusion
Description: In order to compare the total amount of blood transfusion, mean units of blood transfusion was used.
Time Frame: day 3
Population: intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: Mean units of blood transfusion
Arm/Group | Rabeprazole Sodium | Omeprazole
Number analyzed (Participants) | 54 | 52
Mean units of blood transfusion | 1.3 (1.4) | 1.4 (1.3)
Statistical Analysis 1: Comparison: Rabeprazole Sodium vs Omeprazole; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

6. Other Pre Specified Outcome: Duration of Hospital Stay
Time Frame: 6wk
Population: intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Rabeprazole Sodium | Omeprazole
Number analyzed (Participants) | 54 | 52
days | 8.0 (5.6) | 6.7 (2.1)
Statistical Analysis 1: Comparison: Rabeprazole Sodium vs Omeprazole; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: week 6
Arm/Group | Rabeprazole Sodium | Omeprazole
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/52
Other Adverse Events (participants affected / at risk) | 2/54 | 2/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rabeprazole Sodium (N=54) | Omeprazole (N=52)
hepatic enzyme elevation (Hepatobiliary disorders) | 1 (1) | 1 (1)
tonic seizure like activity (Nervous system disorders) | 1 (1) | 0 (0)
Ventricular premature beats (Cardiac disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This was the two-center study and was stopped before the complete enrollment leading to small numbers of subjects statistically underpowered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No